CLINICAL TRIAL: NCT03566563
Title: Epidemiology of Chronic Hepatitis C and Modelling for Disease Burden Study
Brief Title: Epidemiology of Chronic Hepatitis C and Disease Modelling
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2804
Record Dates: First submitted 2018-05-08; First posted 2018-06-25 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C
Keywords: Community Screening; Halfway house; People who inject drugs; Substance users; Released prisoners
MeSH Terms: conditions — Hepatitis C | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ex-Drug Users: These are ex drug users residing at halfway houses
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Patients tested positive for Hepatitis C will be referred to Hospital through the conventional health care services and by an alternative direct access method to determine if this improves linkage to care
  Other Names: Models of Care

SUMMARY:
Hepatitis C (HCV) is a major health problem amongst people who inject drugs (PWID) and have limited contact with health care services. Halfway houses (HH) serve to reintegrate former drug users into society. Strategies to eliminate HCV must focus on screening for HCV amongst HH. Linkage to care for PWID population is an issue globally.

The aim is to determine the sero-prevalence, demographics, disease distribution and factors associated with the risk of HCV transmission amongst former drug users at Halfway Houses. The secondary aim would be to determine the best models of care that can be used to link these individuals to existing healthcare services in a pragmatic, randomised fashion

Halfway Houses are invited to participate in a program of HCV education, point-of-care screening using Oraquick test and staging with Fibroscan® by a small mobile team of healthcare workers. A detailed survey regarding illicit drug injecting practices is performed. Those who are tested positive are referred to medical care.

It is anticipated that the prevalence of Hepatitis C within the drug injecting population along with the stages of liver disease such that models for disease burden can be determined.

DETAILED DESCRIPTION:
This is a pragmatic observational study of point of care HCV screening in the halfway house resident /PWID population.

In the secondary aim the HCV positive subjects are randomised to traditional referral pathway (HCV positive cases attend primary care facilities to get referral to specialist clinic in hospital) and 'direct' open access where the HCV positive cases has direct open access to specialist clinic as above (by passing primary care physicians). We observe the no. of subjects being linkage to specialist care, and HCV treatment

ELIGIBILITY:
Inclusion Criteria:

* Former Drug Users residing in Halfway Houses

Exclusion Criteria:

* Age below 21 years
* Residents of Halfway Houses who have never used drugs

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Halfway House (HH) residents are largely former injecting drug users who have a high prevalence of Hepatitis C. Typically upon release from prisons, there are housed at HH as an interim step prior to re-integration back into society. The prevalence of Hepatitis C within this community allows the estimation of the national prevalence of Hepatitis C in the country.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
HCV Sero-prevalence at Halfway Houses | 24 months
  The number of HCV Sero positive cases at Halfway Houses will be measured

SECONDARY OUTCOMES:
Linkage to Care | 24 months
  The number of patients linked to care will be compared between the intervention arm and conventional arm

OTHER OUTCOMES:
Disease burden estimation | 24 months
  The number of HCV positive cases in Singapore will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Prem H Thurairajah, PhD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No